CLINICAL TRIAL: NCT00891540
Title: Lokal Infiltrations Analgesi Med Ropivakain 0,5 % Versus Ropivakain 0,2 % Versus Placebo Efter Sectio Caesarea: et Prospektivt, Dobbeltblindet, Placebokontrolleret Studie.
Brief Title: Local Infiltration Analgesia With Ropivacaine Versus Placebo in Caesarean Section
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Billy B. Kristensen, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: H-C-2009-019
Record Dates: First submitted 2009-04-30; First posted 2009-05-01 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2009-04

CONDITIONS: Pain, Postoperative; Postoperative Nausea and Vomiting; Cesarean Section
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Local infiltration with Ropivacaine
  Interventions: Drug: Ropivacaine
- 2 (Active Comparator): Local infiltration with Ropivacaine
  Interventions: Drug: Ropivacaine
- 3 (Placebo Comparator): Local infiltration with NaCl
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Ropivacaine — Ropivacaine 0.5%
  Arms: 1
Drug: Ropivacaine — Ropivacaine 0.2%
  Arms: 2
Drug: placebo — Isotonic NaCl
  Arms: 3

SUMMARY:
The purpose of this study is to compare systematic local infiltration with Ropivacaine 0.5 % versus Ropivacaine 0.2 % versus Placebo in patients undergoing elective caesarean section.

The hypothesis is that systemic local infiltration will reduce pain and postoperative opioid consumption.

ELIGIBILITY:
Inclusion Criteria:

* eligible for elective caesarean section
* able to speak and understand Danish
* able to give informed consent

Exclusion Criteria:

* alcohol or medical abuse
* allergies to local anesthetics
* age < 18 years
* intolerance to opioids

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | 24 hours

SECONDARY OUTCOMES:
Postoperative nausea and vomiting (PONV) | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre University Hospital, Copenhagen, Hvidovre, Denmark